CLINICAL TRIAL: NCT06489314
Title: A Brief, Task-shifted Treatment to Improve Father Depression and Child Outcomes in Kenya: A Pilot Effectiveness-implementation Trial
Brief Title: Mental Health Treatment to Improve Father Depression and Child Outcomes in Kenya
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Moi Teaching and Referral Hospital (Other)
Responsible Party: Principal Investigator, Ali Giusto, PhD, Assistant Professor, Florida International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1K23MH128742-01A1 (NIH)
Record Dates: First submitted 2024-06-25; First posted 2024-07-05 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-04

CONDITIONS: Father-Child Relations; Depression; Alcohol Use, Unspecified
Keywords: Randomized Control Trial; Hybrid-Type 1 Trial; Depression; Alcohol Use; Peer Counseling; Task-Shifting; Fathers; Youth Mental Health; Kenya
MeSH Terms: conditions — Depression; Alcohol Drinking | interventions — Lead; Educational Status; alpha 1-Antichymotrypsin

STUDY DESIGN:
Intervention Model Description: Hybrid type-1 waitlist control pilot trial. Fathers at risk for depression will be randomized randomized 2:1 to the intervention or waitlist. All participants will receive referrals to treatment at usual at baseline. Waitlist participants will be offered the intervention at the completion of their assessments.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEAD Intervention (Experimental): LEAD consists of behavioral activation (BA) and motivational interviewing (MI), as well as discussions of masculinity and a family focus throughout to target father's depression symptoms and common comorbidities, like drinking. LEAD is guided by a manual (in Swahili and English). It includes five, 60-90-minute weekly sessions. LEAD was adapted for context based on formative work. Each session begins with MH assessment and review of activity completion and ends with homework to monitor activities. LEAD uses MI strategies to engage men in the treatment and increase commitment to addressing problems. MI strategies are then integrated throughout. (Session 1-5) to enhance father motivation to complete activities as well as to build self-efficacy (e.g., when reviewing homework, peer-father counselors reflect successes).
  Interventions: Behavioral: LEAD (Learn, Engage, Act, Dedicate)
- Waitlist Control (No Intervention): Those randomized to WL will complete assessments and be monitored at each timepoint; they will be offered LEAD following the last assessment. In a pilot, a control allows for a realistic examination of recruitment, randomization, implementation of LEAD, assessment procedures, and retention. If safety concerns arise, referrals and safety procedures will be implemented.

INTERVENTIONS:
Behavioral: LEAD (Learn, Engage, Act, Dedicate) — LEAD is a 5-session behavioral activation (BA) intervention delivered by peer-father counselors. LEAD also incorporates motivational interviewing (MI) and masculinity discussion strategies. This is a task-shifted intervention meaning mental health service tasks are delegated to non-specialist providers, in this case peer-fathers, as opposed to a specialized workforce (e.g., psychiatrists, psychologists).
  Arms: LEAD Intervention

SUMMARY:
The goal of this study is to evaluate the feasibility and acceptability of a peer-father counselor delivered psychosocial intervention for fathers at risk for depression and some alcohol use in Eldoret, Kenya in a pilot randomized control trial (RCT). The study draws on existing partnerships with Moi Teaching and Referral Hospital (MTRH) and AMPATH (a consortium of North American and Kenyan institution conducting research) in Kenya. It will also build on already completed preliminary work with AMPATH/MTRH that showed proof-of-concept for 'Learn, Engage, Act, Dedicate' (LEAD), a 5-session task-shifted psychosocial intervention for fathers in Eldoret, Kenya. Proof-of-concept findings with nine fathers and families were promising with high participant satisfaction and improvements in father depression, alcohol use, parenting, and child mental health. This supported pursuit of a pilot RCT, proposed here, to explore preliminary effectiveness of LEAD and its implementation. Specifically, investigators aim to conduct a pilot RCT with fathers (n=102) randomized to either LEAD or a waitlist control group (with treatment offered at the end of the waitlist period) to explore change in fathers' mental health (MH); explore drivers of change in father MH, father parenting, and child MH (or non-response); and explore the feasibility and acceptability of implementing a peer-father counselor delivered MH treatment for fathers. Investigators will also refer all participants that screen positive for depression and alcohol use problems at recruitment (the WL control and intervention group) to services in the area using existing referral to care procedures.

DETAILED DESCRIPTION:
Investigators will conduct a pilot randomized control trial using an implementation-effectiveness Hybrid Type I design. Fathers with depression (n=102) will be randomized to depression treatment LEAD or a wait list (WL) control at a rate of 2:1. LEAD will be offered to the WLC following treatment. This is a pilot. Aims focus on preliminary indicators of effectiveness and feasibility and acceptability (implementation). Data will inform a larger trial.

The objective of this study is to conduct a pilot randomized control trial using an implementation-effectiveness Hybrid Type I design to explore improvements in father depression using a brief, task-shifted intervention and explore implementation feasibility and acceptability. Participants will be randomized to LEAD (Learn, Act, Engage, Dedicate), a 5-session behavioral activation and motivational interviewing treatment, or to a waitlist control group (WL) in Eldoret, Kenya among men with depression symptoms (WL participants will be offered treatment at their final assessment). Fathers (n=102) will be randomized to treatment at a rate of 2:1; assessments will occur at baseline, post treatment, and 1 and 3 months post. As part of Aim 1, investigators will explore changes between groups in father depression post-treatment as measured by the PHQ-9, as well as secondary outcomes of drinking, parenting, interparental problems, and child mental health assessed among men, a co-caregiver, and one child with surveys (Women (n=102) and children (n=102) will only report on themselves and family outcomes not father mental health). The WL will receive all assessments at each timepoint and be monitored for safety; rates of attrition will be tracked throughout as well as rates of those possibly pursuing care during the trial. Next, investigators will explore potential mechanisms of change on father depression and family and child outcomes using survey measures as well as qualitative data - both semi-structured interviews 1 month post with men and family participants (n=30) and transcript analysis (n=20) of men and families showing different patterns of response or non-response. Lastly, investigators will explore implementation feasibility and acceptability as measured by qualitative interviews assessing acceptability and barriers/facilitators to delivery, including social determinant barriers such as economic hardship, and brief surveys with providers 1-month after treatment, as well as fidelity (adherence to intervention steps), coded from 20% of randomly selected session transcripts based on a previously developed and piloted adherence tool, and participant retention and attendance.

ELIGIBILITY:
Inclusion Criteria:

1. Male between the ages of 18-65;
2. Live with and be responsible for at least one child between the ages of 8 and 17 years of age;
3. Screen positive for depression symptoms, operationalized as a score above 5 on the patient health questionnaire (PHQ-9);
4. Any reported alcohol use in the past 45 days measures with the AUDIT (score 1 or above);
5. Child at risk of mental health issues as indicated by a score above 13 on the Strengths and Difficulties Questionnaire (SDQ) reported on by any caregiver;
6. Willingness for co-caregiver and target child to participate in assessments (previously piloted strategy).

Exclusion Criteria:

1. Severe depression symptoms indicated a score above 19 on the PHQ-9;
2. Severe risk/likely alcohol dependence that warrants medical management indicated as a score 20 or above on the alcohol use disorder identification test (AUDIT);
3. Violent legal offenses (one question);
4. Indicators of severe violence at home assessed with key items from the Conflict Tactics Scale (CTS), following previously used criteria. If any couple member answers yes (related to the father) to either of the following items: "punched or hit my partner with something that could hurt" and "kicked my partner," couples will be excluded. Couple members who answer yes to any of the following items: "I/he used a knife or gun on my partner/me," "I/he choked my partner/me," "I/he slammed my partner/me against a wall," "I/he beat up my partner/me," "I/he burned or scalded my partner/me on purpose," will be excluded.
5. Inability to provide informed consent of complete procedures in Swahili or English;
6. serious mental illness (current or history).
7. Youth in age range not at risk for MH problems: No Score <13 to 40 on the SDQ as reported by both caregivers

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Fathers
Enrollment: 116 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Depression Symptoms | Baseline (Time point 1, in year 1); 6-10 weeks after baseline; 10-14 weeks after baseline; 19-23 weeks after baseline
  Patient Health Questionnaire (PHQ-9): a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression, previously validated and used in Kenya.

SECONDARY OUTCOMES:
Type of Alcohol Use | Baseline (Time point 1, in year 1); 6-10 weeks after baseline; 10-14 weeks after baseline; 19-23 weeks after baseline
  AUDIT (Alcohol Use Disorders Identification Test): a simple and effective method of screening for unhealthy alcohol use, defined as risky or hazardous consumption or any alcohol use disorder. The AUDIT has been has been previously validated in Kenya.
Gender Norms | Baseline (Time point 1, in year 1); 6-10 weeks after baseline; 10-14 weeks after baseline; 19-23 weeks after baseline
  Gender-Equitable Men (GEM) Scale: assesses men's beliefs about gender norms and gender roles. Higher scores correspond with more equitable gender views. This scale has been previously used in Kenya to measure inequitable attitudes
Disrupted Parenting | Baseline (Time point 1, in year 1); 6-10 weeks after baseline; 10-14 weeks after baseline; 19-23 weeks after baseline
  Alabama Parenting Questionnaire (APQ - Father Involvement Scale) (Adapted): The involvement subscale of the Alabama Parenting Questionnaire (APQ) assesses father level of participation in their child's life, such as father attendance at child activities or help with homework. Items have been adapted to enhance local acceptability, understandability, and completeness with minor adaptations and previously piloted in Eldoret, Kenya.
Interparental Problems | Baseline (Time point 1, in year 1); 6-10 weeks after baseline; 10-14 weeks after baseline; 19-23 weeks after baseline
  Family Togetherness Scale (FTS): Interparental problems will be assessed with 25 items, such as "How often does your family have quarrels?" Items relate to issues of family structure, couple emotional climate, and couple communication. These items were locally developed (Puffer et al., 2018), and have been validated in the context. Scores are averaged by reporter (men reliability = 0.95; co-caregivers reliability = 0.96; Child reliability = 0.95), with higher scores indicating poorer family functioning in this study.
Child Mental Health | Baseline (Time point 1, in year 1); 6-10 weeks after baseline; 10-14 weeks after baseline; 19-23 weeks after baseline
  Strengths and Difficulties Questionnaire (SDQ): The Strengths and Difficulties Questionnaire (SDQ) is a 25 item brief youth mental health screening questionnaire relevant to 3 to 17 year olds that has been validated for both caregiver and youth report. The measures assesses emotional symptoms (5 items); 2) conduct problems (5 items) ; 3) hyperactivity/inattention (5 items) ; 4) peer relationship problems (5 items); 5) prosocial behavior (5 items), as well as a total score (20 items. We will use the total item score. The SDQ has previously used in Kenya and Eldoret with good performance.

OTHER OUTCOMES:
Treatment Engagement | through the treatment period, 2- 8 weeks after baseline
  engagement is defined as the percent of participant attendance these are sessions attended as scheduled or rescheduled. This will be tracked and logged by RA during treatment.
Activity Completion | through the treatment period, 2- 8 weeks after baseline
  RA's will code participants activity schedules that they complete as part of their treatment homework. Homework consists of scheduling activities that are pleasant, healthy or aligned with values. Schedules will be coded as the the percentage of positive activities they indicted that they would complete in the previous session as well as the frequency activities completed.
Positive Emotional Reinforcement | through the treatment period, 2- 8 weeks after baseline
  Positive emotion or positive reinforcement following activity completion will be assessed through the activities schedules completed as part of intervention homework. When reviewing homework in session, patient and counselor will discuss and write down the emotion felt after completing a scheduled activity. These schedules will coded by RA's following each treatment session for patient's report of what activities they completed and the emotion felt immediately after the completed activity. Emotions will be coded as 'positive' (e.g., proud, relief, mastery, pleasurable) or 'not positive' (e.g., boring, angry, frustrated) resulting in the percentage of positive emotion of completed activities.
Fidelity Checklist | through the treatment period, 2- 8 weeks after baseline
  All intervention sessions will be audiotaped; 20 percent of tapes will be transcribed, translated to English, and then reviewed by the PI and project coordinator. Fidelity ratings will be based on a previously piloted assessment of adherence and competency. A "fidelity score" will be calculated based on the proportion of key intervention components delivered as intended across sessions (Yes/No) as well as quality of delivery (1-4, 4 excellent).
Retention | through the treatment period, 2- 8 weeks after baseline
  retention will be analyzed as the percentage of fathers: attending one session or more session, attending 75 percent of session or more, and those who dropped out of LEAD
Participation | through the treatment period, 2- 8 weeks after baseline
  analyzed as the percentage of fathers who enroll in LEAD who are eligible and percent excluded due to ineligibility
Feasibility of the Intervention and Implementation | 6-10 weeks after baseline
  4-item feasibility of intervention measure. Scale 1-5 completely disagree to completely agree.
Acceptability (quantitative) | 6-10 weeks after baseline
  4-item acceptability of intervention measure. Scale 1-5 completely disagree to completely agree.
Appropriateness | 6-10 weeks after baseline
  4-item measures assessing intervention appropriateness . Scale 1-5 completely disagree to completely agree.
General Counseling Competency | through the treatment period, 2- 8 weeks after baseline
  General clinical competency will be coded and rated using a previously adapted and piloted version of the ENhancing Assessment of Common Therapeutic factors (ENACT) rating scale using session recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Giusto, PhD, Principal Investigator — Florida International University
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: Undecided
This will be dependent on what partners in Kenya prefer.

REFERENCES:
- [Background] Monahan PO, Shacham E, Reece M, Kroenke K, Ong'or WO, Omollo O, Yebei VN, Ojwang C. Validity/reliability of PHQ-9 and PHQ-2 depression scales among adults living with HIV/AIDS in western Kenya. J Gen Intern Med. 2009 Feb;24(2):189-97. doi: 10.1007/s11606-008-0846-z. Epub 2008 Nov 20. PMID 19031037
- [Background] Puffer ES, Healy EF, Green EP, Giusto AM, Kaiser BN, Patel P, Ayuku D. Family Functioning and Mental Health Changes Following a Family Therapy Intervention in Kenya: a Pilot Trial. J Child Fam Stud. 2020 Dec;29(12):3493-3508. doi: 10.1007/s10826-020-01816-z. Epub 2020 Sep 24. PMID 33664559
- [Background] Puffer ES, Giusto A, Rieder AD, Friis-Healy E, Ayuku D, Green EP. Development of the Family Togetherness Scale: A Mixed-Methods Validation Study in Kenya. Front Psychol. 2021 Jun 8;12:662991. doi: 10.3389/fpsyg.2021.662991. eCollection 2021. PMID 34168594
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Vreeman RC, Scanlon ML, Marete I, Mwangi A, Inui TS, McAteer CI, Nyandiko WM. Characteristics of HIV-infected adolescents enrolled in a disclosure intervention trial in western Kenya. AIDS Care. 2015;27 Suppl 1(sup1):6-17. doi: 10.1080/09540121.2015.1026307. PMID 26616121
- [Background] Babor, T. F., Higgins-Biddle, J. C., Saunders, J. B. & Monteiro, M. G. Audit. The Alcohol Use Disorders Identification Test (AUDIT): guidelines for use in primary care (2001)
- [Background] Pulerwitz, J. & Barker, G. Measuring Attitudes toward Gender Norms among Young Men in Brazil: Development and Psychometric Evaluation of the GEM Scale. Men and Masculinities 10, 322-338 (2007).
- [Background] Essau, C. A., Sasagawa, S. & Frick, P. J. Psychometric properties of the Alabama parenting questionnaire. Journal of Child and Family Studies 15, 595-614 (2006).
- [Background] Kohrt BA, Jordans MJ, Rai S, Shrestha P, Luitel NP, Ramaiya MK, Singla DR, Patel V. Therapist competence in global mental health: Development of the ENhancing Assessment of Common Therapeutic factors (ENACT) rating scale. Behav Res Ther. 2015 Jun;69:11-21. doi: 10.1016/j.brat.2015.03.009. Epub 2015 Mar 24. PMID 25847276
- [Derived] Giusto A, Jaguga F, Aburi D, Korir M, Maina W, Rono W, Greenlee M. Protocol for a Hybrid-type 1 pilot study of a randomized control trial of a brief, peer-delivered treatment to improve father depression and child mental health in Kenya. PLoS One. 2025 Jun 26;20(6):e0325902. doi: 10.1371/journal.pone.0325902. eCollection 2025. PMID 40570024